CLINICAL TRIAL: NCT03238222
Title: A Brief Physiotherapist-led Behaviour Change Intervention to Facilitate Walking in Older People With Peripheral Arterial Disease: a Randomised Controlled Trial
Brief Title: Motivating Structured Walking Activity in Intermittent Claudication
Acronym: MOSAIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); The Dunhill Medical Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17/LO/0568; R477/0516 (Other Grant/Funding Number: Dunhill Medical Trust)
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Disease
Keywords: Walking; Six-Minute Walk Distance; Illness Perceptions; Theory of Planned Behaviour
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases | interventions — Mosaicism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOSAIC Treatment (Experimental): MOSAIC treatment plus Usual NHS Care. MOSAIC treatment comprises 2 x 60-minute individual face-to-face consultations (weeks 1 & 2) and 2 x 20-minute follow-up telephone calls (weeks 6 & 12) with a trained physiotherapist.
  Interventions: Behavioral: MOSAIC
- Usual Care Comparison (No Intervention): Usual NHS care for people with intermittent claudication typically consists of an initial assessment, drug therapy and simple advice to walk provided by a vascular specialist and delivered in the vascular outpatient clinic.

INTERVENTIONS:
Behavioral: MOSAIC — MOSAIC comprises 2 x 60-minute individual face-to-face consultations (weeks 1 & 2) and 2 x 20-minute follow-up telephone calls (weeks 6 & 12) delivered at a convenient time and location of participant's choice (local NHS Trust or participant's home). All sessions are delivered by a trained Band 6/7 physiotherapist. All participants randomized to receive MOSAIC will be provided with a pedometer and a patient manual which will include information on intermittent claudication, risk factors, walking guidelines, goal setting, problem solving and action planning worksheets and a walking diary.
  Other Names: Motivating Structured walking Activity in IC
  Arms: MOSAIC Treatment

SUMMARY:
Peripheral arterial disease can cause leg pain or discomfort (called intermittent claudication (IC)), which limits the ability to walk and carry out everyday activities. Lifestyle changes, like increasing walking, can lead to improvements, but can be a challenge to begin and then continue. The aim of this study is to investigate if a physiotherapist-led, behaviour change treatment effects walking in people with IC. The treatment is designed to build an understanding of IC and walking exercise and help individuals develop strategies to increase regular walking. The trial will recruit 192 adults (aged 50 years and over) with IC. All participants will visit King's College London or their local hospital to complete two short walking tests and answer questionnaires about their daily activities, beliefs about their symptoms and treatment, quality of life and the costs of having IC.

Participants will then be randomly assigned to receive either the new treatment or continue with their usual NHS care. The new treatment involves two 60-minute face-to-face sessions (at the participant's home or local hospital) and two 20-minute telephone calls with a physiotherapist who will discuss participants' understanding and beliefs about IC, walking and help participants to set goals and plans to increase walking over 12 weeks. Participants will be provided with a step counter (pedometer) and walking record.

After 12 weeks, all participants will attend a second appointment where they will repeat the walking tests and fill out another set of questionnaires. A final set of questionnaires will be completed by all participants after 6 months (by post or electronically). Some participants will be invited to provide feedback on their experience of the treatment and trial by telephone or a face-to-face interview with a researcher.

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years of age;
* established PAD (Ankle Brachial Pressure Index ≤0.90 and/or radiographic evidence or clinician reported diagnosis) and IC (presence of symptoms reported on the San Diego Claudication Questionnaire)
* able to participate in MOSAIC
* able and willing to provide informed consent

Exclusion Criteria:

* Unstable IC (self-reported change in symptoms during previous 3 months)
* walking >90 minutes/week (reported on Brief International Physical Activity Questionnaire
* contraindications to walking exercise (e.g., unstable angina) confirmed by their vascular specialist
* have completed any prescribed supervised exercise sessions in the previous 6 months or been offered prescribed exercise sessions in the next 6 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-11-09 (Estimated); Study Completion 2021-01-09 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Distance | 3 months
  6 Minute Walking Distance (in metres) measured during a self-paced, standardised 6 Minute Walk Test conducted around a level, 100-foot circuit.

SECONDARY OUTCOMES:
6 Minute Walk Distance (6MWD) | Baseline and 3 months
  6 Minute Walking Distance (in metres) measured during a self-paced, standardised 6 Minute Walk Test conducted around a level, 100-foot circuit.
Self-reported Maximum Walking Distance | Baseline, 3 and 6 months
  Single global item
Self-Reported Walking Ability | Baseline, 3 and 6 months
  Walking Estimated-Limitation Calculated by History (WELCH)
Activities of Daily Living | Baseline, 3 and 6 months
  Nottingham Extended Activities of Daily Living (NEADL)
Health-Related Quality of Life | Baseline, 3 and 6 months
  Vascular Quality of Life Questionnaire-6 (VascuQol-6)

OTHER OUTCOMES:
Treatment Cognitions | Baseline, 3 and 6 months
  Theory of Planned Behaviour Questionnaire
Illness Cognitions | Baseline, 3 and 6 months
  Brief Illness Perceptions Questionnaire (BIPQ)
Walking Adherence | Baseline, 3 and 6 months
  Exercise Adherence Rating Scale
Resource Use | Baseline, 3 and 6 months
  Client Service Receipt Inventory
Health Related Quality of Life | Baseline, 3 and 6 months
  Euroqol- 5D-5L
Pain Free Walking Ability | Baseline and 3 months
  Patient-reported pain free walking time (seconds) and distance (metres) during the 6 Minute Walk Test
Maximal Walking Ability | Baseline and 3 months
  The maximum time (seconds) and distance (metres) walked before stopping during a 6 Minute Walk Test

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Patel, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (9):
- United Kingdom (9):
  - Dartford and Gravesham NHS Trust (GSTT PIC site), Dartford, Kent
  - Maidstone and Tunbridge Wells NHS Trust (GSTT PIC site), Maidstone, Kent
  - Ashford & St Peter's NHS Foundation Trust, Ashford, Surrey
  - Guy's & St Thomas NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Lewisham and Greenwich NHS Trust (GSTT PIC site), London
  - Royal Free London NHS Foundation Trust, London
  - St George's University Hospital NHS Foundation Trust, London
  - The Royal London Hospital, Barts Heatth NHS Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bearne LM, Volkmer B, Peacock J, Sekhon M, Fisher G, Galea Holmes MN, Douiri A, Amirova A, Farran D, Quirke-McFarlane S, Modarai B, Sackley C, Weinman J, Bieles J; MOSAIC Trial Collaboration. Effect of a Home-Based, Walking Exercise Behavior Change Intervention vs Usual Care on Walking in Adults With Peripheral Artery Disease: The MOSAIC Randomized Clinical Trial. JAMA. 2022 Apr 12;327(14):1344-1355. doi: 10.1001/jama.2022.3391. PMID 35412564